CLINICAL TRIAL: NCT01618656
Title: FAAH-Inhibitor for Cannabis Dependence
Brief Title: Safety and Efficacy of a FAAH-Inhibitor to Treat Cannabis Withdrawal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1202009714; U01DA033267 (NIH)
Record Dates: First submitted 2012-06-05; First posted 2012-06-13 (Estimated); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-01

CONDITIONS: Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-04457845 (Active Comparator): 2/3 of subjects will be randomized to fatty acid amide hydrolase (FAAH) inhibitor 4mg
  Interventions: Drug: PF-04457845
- Placebo (sugar pill) (Placebo Comparator): 1/3 of subjects will be randomized to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04457845 — Study medication will be administered at 4mg by mouth daily for four weeks.
  Arms: PF-04457845
Drug: Placebo — Sugar pill
  Arms: Placebo (sugar pill)

SUMMARY:
Cannabis dependence is associated with changes in the brain's cannabinoid system. When cannabis dependent individuals try to quit using cannabis, some of them experience problems that make it difficult for them to achieve and maintain abstinence. Therefore, reducing the problems related to quitting cannabis may facilitate abstinence. One way to do this is by harnessing the brain's capacity to make its own cannabis-like substances - endocannabinoids. One of the main endocannabinoids is anandamide. The study is based on the hypothesis that the problems related to quitting cannabis use will be reduced by increasing the brain levels of anandamide. Furthermore, by reducing the problems related to quitting cannabis, people will be less likely to relapse. Brain anandamide levels will be increased by blocking the breakdown of anandamide using a fatty acid amide hydrolase inhibitor (FAAH-I). The effects of a novel FAAH-I cannabis withdrawal and relapse in cannabis dependent subjects will be studied in a double-blind, randomized, controlled, proof-of-concept study. Cannabis-dependent subjects will receive placebo or the FAAH-inhibitor PF-04457845 in a 2:1 randomization. The trial consists of a 1 week inpatient stay to achieve abstinence, a 3 week outpatient treatment phase. Cannabis withdrawal will be measured during the inpatient phase. Cannabis use and urinary THC-COOH levels will be measured during the entire study. The treatment phase will be followed by a safety follow up phase of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Ages 18-55 (inclusive)
3. Cannabis Dependence

Exclusion Criteria:

1. Allergies or intolerance to FAAH-Inhibitors
2. Current significant medical or other comorbidities

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-09-12 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2016-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] D'Souza DC, Cortes-Briones J, Creatura G, Bluez G, Thurnauer H, Deaso E, Bielen K, Surti T, Radhakrishnan R, Gupta A, Gupta S, Cahill J, Sherif MA, Makriyannis A, Morgan PT, Ranganathan M, Skosnik PD. Efficacy and safety of a fatty acid amide hydrolase inhibitor (PF-04457845) in the treatment of cannabis withdrawal and dependence in men: a double-blind, placebo-controlled, parallel group, phase 2a single-site randomised controlled trial. Lancet Psychiatry. 2019 Jan;6(1):35-45. doi: 10.1016/S2215-0366(18)30427-9. Epub 2018 Dec 6. PMID 30528676

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04457845 (4mg by Mouth Daily for 4 Weeks): 2/3 of subjects will be randomized to fatty acid amide hydrolase (FAAH) inhibitor 4mg
  PF-04457845: Study medication will be administered at 4mg by mouth daily for four weeks.
- Placebo (Sugar Pill, by Mouth Daily for 4 Weeks): 1/3 of subjects will be randomized to placebo
  Placebo: Sugar pill
Period: Overall Study
Arm/Group | PF-04457845 (4mg by Mouth Daily for 4 Weeks) | Placebo (Sugar Pill, by Mouth Daily for 4 Weeks)
Started | 46 | 24
Completed | 38 | 20
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04457845 (4mg by Mouth Daily for 4 Weeks) | Placebo (Sugar Pill, by Mouth Daily for 4 Weeks) | Total
Number analyzed (Participants) | 46 | 24 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 24 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 46 | 24 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 39 | 20 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 12 | 36
  White | 18 | 9 | 27
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 24 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Marijuana Withdrawal Checklist (MWC)
Description: 32-item checklist evaluating potential symptoms of cannabis withdrawal, lower values reflect lesser severity of withdrawal symptoms (lower scores represent a better outcome).
  Min: 0 Max: 96
Time Frame: The MWC was administered on Day 0, Day 1, Day 2, Day 3, and Day 4 (during the inpatient phase when withdrawal peaks) to assess change from baseline (Day 0). The scores from each time point and subject were calculated to report the mean score for each arm.
Population: Missing data and the removal of outliers led to differences between the total number of participants and the sample for this variable
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PF-04457845 (4mg by Mouth Daily for 4 Weeks) | Placebo (Sugar Pill, by Mouth Daily for 4 Weeks)
Number analyzed (Participants) | 31 | 19
score on a scale | 6.04 [4.43 to 8.24] | 11 [7.78 to 15.57]

2. Primary Outcome: Change in Self Reported Cannabis Use at the End of 4 Weeks
Description: Subject quantifies and reports frequency of cannabis use prior to study participation and during the 4 week period. Lower scores reflect less cannabis usage, while higher scores reflect more frequent usage.
  Min: 0 Max: undeterminable, varies per patient and their usage.
Time Frame: Administered weekly for 4 weeks to assess change from baseline (Day 0). The scores from each time point and subject were calculated to report the mean score for each arm.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: joints per day
Arm/Group | PF-04457845 (4mg by Mouth Daily for 4 Weeks) | Placebo (Sugar Pill, by Mouth Daily for 4 Weeks)
Number analyzed (Participants) | 32 | 19
joints per day | 0.40 [0.25 to 0.62] | 1.27 [0.82 to 1.97]

3. Primary Outcome: Change in THC-COOH Quantification at the End of 4 Weeks
Description: Subjects provide urine samples to quantify levels of THC.
Time Frame: Samples obtained weekly for 4 weeks to assess change from baseline (Day 0). The results from each time point and subject were calculated to report the mean score for each arm.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | PF-04457845 (4mg by Mouth Daily for 4 Weeks) | Placebo (Sugar Pill, by Mouth Daily for 4 Weeks)
Number analyzed (Participants) | 31 | 19
ng/mL | 265.55 [175.60 to 401.57] | 657.92 [381.60 to 1134.30]

4. Secondary Outcome: Change in Polysomnography
Description: Polysomnography (PSG) is a comprehensive reading of biophysiological changes that occur during sleep, including identification of sleep stage. A mean and standard deviation of their data points during sleep stages were calculated to determine change from baseline to the end of study treatment.
Time Frame: Polysomnography was collected two nights prior to baseline visit, for three nights during study treatment and two nights after four weeks of study treatment. A mean was calculated to assess change from baseline (Day 0).
Population: The units analyzed reflects the number of data points (sum of participants per drug condition across time) was 42 in the placebo group and 82 in the PF-04457845 group.
  Missing data and the removal of outliers led to differences between the total number of participants and the sample for this variable.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Number of Data Points
Arm/Group | PF-04457845 (4mg by Mouth Daily for 4 Weeks) | Placebo (Sugar Pill, by Mouth Daily for 4 Weeks)
Number analyzed (Participants) | 31 | 19
Number analyzed (Number of Data Points) | 82 | 42
minutes | 89.56 (35.20) | 69.29 (27)

5. Other Pre Specified Outcome: Feeling States
Description: Visual analog scale for feeling states (depression, anxiety, irritability)
Time Frame: Administered on Day 0, Day 1, Day 2, Day 3, and Day 4 (Once pre-treatment and during the inpatient phase 'acute abstinence') to assess change from baseline (Day 0)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Plasma Endocannabinoid Levels
Description: Measurement of circulating plasma Anandamide
Time Frame: Samples obtained at the following study visits: Day -1, Day 0, Day 2, Day 4, Week 2, Week 3, Week 4 to assess change from baseline (Day 0)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | PF-04457845 (4mg by Mouth Daily for 4 Weeks) | Placebo (Sugar Pill, by Mouth Daily for 4 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/24
Other Adverse Events (participants affected / at risk) | 31/46 | 14/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-04457845 (4mg by Mouth Daily for 4 Weeks) (N=46) | Placebo (Sugar Pill, by Mouth Daily for 4 Weeks) (N=24)
Headache (Nervous system disorders) | 7 (12) | 5 (8)
Trouble Concentrating (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stuffy Nose (General disorders) | 2 (2) | 2 (2)
Sneezing (General disorders) | 1 (1) | 1 (1)
Fluid Filled Cyst on Left Wrist (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chest Congestion (General disorders) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Red Marks/Skin Irritation at PSG Electrode Placement (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash from Tape used for PSG Electrode Application (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eye Twitch (Eye disorders) | 0 (0) | 1 (1)
Lightheaded after Blood Draw (Nervous system disorders) | 1 (1) | 1 (1)
Right Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Loose Stool (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric Paralysis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
High Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Syncopal Episode (Related to Phlebotomy) (Nervous system disorders) | 0 (0) | 1 (1)
Sleep Disturbances (Nervous system disorders) | 0 (0) | 1 (1)
Itchy Throat (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Fever (General disorders) | 2 (2) | 1 (1)
Jammed Pinky Finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Feet Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Scratched Cornea (Eye disorders) | 1 (1) | 0 (0)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Sharp Rib Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pressure in Head (Nervous system disorders) | 1 (1) | 0 (0)
Sinus Pressure (General disorders) | 1 (1) | 0 (0)
Tooth Pain (General disorders) | 1 (1) | 0 (0)
Muscle Strain in Back (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Runny Nose (General disorders) | 2 (2) | 0 (0)
Itchy Throat (General disorders) | 1 (1) | 0 (0)
Sore Throat (General disorders) | 4 (4) | 0 (0)
Dry Skin on Face (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Foot Laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cyst Under Eye (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swollen Lymph Node in Groin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lyme Disease (Nervous system disorders) | 1 (1) | 0 (0)
Chest Tightness (General disorders) | 1 (1) | 0 (0)
Feeling Faint (General disorders) | 1 (1) | 0 (0)
Trouble Sleeping (Nervous system disorders) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 1 (1) | 0 (0)
Ringworm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Low Phosphorus Levels (Vascular disorders) | 1 (1) | 0 (0)
Ear Popping (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Worsening of Existing Hernia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nose Bleed (General disorders) | 1 (1) | 0 (0)
Gas (Gastrointestinal disorders) | 1 (1) | 0 (0)
Burst Blood Vessel in Right Eye (Eye disorders) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sweating (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes